

# **Statistical Analysis Plan Approval**

| Date: | 04Dec2020 |
|-------|--------------|
| То: | Study File |
| From: | Statistician |

**Re:** Statistical Analysis Plan Approval for Study *D5780C00007* 

The Statistical Analysis Plan, version 3.0, for Study D5780C00007 has been reviewed and approved.

| Name:<br>Role: | Statistician | Signatur December 4, 2020 Date: |
|---|---|---|
| Name:<br>Role: | Statistical Programmer | Signature December 8, 2020 Date: |
| Name:<br>Role: | Clinical Development Lead | Signature December 4, 2020 Date: |
| Name:<br>Role: | Early CVRM Biometrics Team<br>Leader | Signature December 4, 2020 Date: |

# **Statistical Analysis Plan**

A Randomized, Placebo controlled Phase 2b Study to Evaluate the Safety and Efficacy of MEDI6012 in Acute ST Elevation Myocardial Infarction

Protocol Number: D5780C00007

# **TABLE OF CONTENTS**

| 1 | INT | RODUCTION6 | |
|---|---|---|---|
| 2 | STU | DY OVERVIEW | 6 |
| | 2.1 | Study Objectives | 6 |
| | | 2.1.1Primary Study Objective(s) | 6 |
| | | 2.1.2Secondary Study Objectives | 6 |
| | | 2.1.3Exploratory Study Objectives | 7 |
| | 2.2 | Study Design | 8 |
| | 2.3 | Treatment Assignment and Blinding | 10 |
| | 2.4 | Sample Size | 11 |
| 3 | STA | TISTICAL METHODS | 11 |
| | 3.1 | General Considerations | 11 |
| | 3.2 | Analysis Populations | 12 |
| | 3.3 | Study Subjects | |
| | | 3.3.1Subject Disposition and Completion Status | |
| | | 3.3.2Demographics and Baseline Characteristics | 13 |
| | | 3.3.3Study Drug Exposure | 13 |
| | | 3.3.4Concomitant Medications | 14 |
| | 3.4 | Efficacy Analyses | |
| | | 3.4.1Primary Efficacy Endpoint(s) and Analyses | |
| | | 3.4.1.1 Primary Efficacy Endpoint(s) | |
| | | 3.4.1.2 Handling of Dropouts and Missing Data | |
| | | 3.4.1.3 Primary Efficacy Analysis | 14 |
| | | 3.4.1.4 Additional Analyses of the Primary Efficacy Endpoint(s) | |
| | | 3.4.1.5 Subgroup Analyses | |
| | | 3.4.2Secondary Efficacy Endpoint(s) and Analyses | |
| | | 3.4.2.1 Secondary Efficacy Endpoint(s) | |
| | | 3.4.2.2 Handling of Dropouts and Missing Data | 16 |
| | | 3.4.2.3 Secondary Efficacy Analyses | |
| | | 3.4.2.4 Subgroup Analyses | |
| | | 3.4.3Other Efficacy Analyses | |
| | 3.5 | Pharmacodynamic Endpoint(s) and Analyses | |
| | | 3.5.1.1 Pharmacodynamic Endpoint(s) | |
| | | 3.5.1.2 Analysis of Pharmacodynamic Endpoint | |
| | 3.6 | Safety Analyses | |
| | | 3.6.1Adverse Events and Serious Adverse Events | |
| | | 3.6.2Adverse Events of Special Interest | |
| | | 3.6.3Deaths and Treatment Discontinuations due to Adverse Events | 20 |

| | | 3.6.4Clinical Laboratory Evaluation | 20 |
|---|---|---|---|
| | | 3.6.4.1 Vital Signs | 20 |
| | | 3.6.4.2 Electrocardiogram | |
| | 3.7 | Immunogenicity | |
| | 3.8 | Pharmacokinetics | |
| | 3.9 | COVID-19 Analyses | |
| 4 | | RIM ANALYSIS | |
| 5 | | RENCES | |
| 6 | | SION HISTORY | |
| Ü | V LICE | | |
| LIST | OF | TABLES | |
| Table | 2.1 | Primary Objective and Associated Endpoint | 6 |
| Table | 2.2 | Secondary Objectives and Associated Endpoints | 6 |
| Table | 2.3 | Exploratory Objectives and Associated Endpoints | 7 |
| Table | | Analysis Populations | |
| Table | 3.2 | Post-randomization Analysis Subgroups | 15 |
| LIST | OF I | FIGURES | |
| Figure | 2.1 | Overall Study Schema | 9 |
| Figure | | Study Flow Diagram for Cohort A: 2-Dose Regimen | |
| Figure | 2.3 | Study Flow Diagram for Cohort B: 6-Dose Regimen | |
| Figure | e 4.1 | Predictive power against observed interim relative infarct size reduction when 30% of the Primary Efficacy Analysis Population is | |
| Figure | . 1 2 | enrolled and complete their final study visit Predictive power against observed interim ejection fraction increase | |
| rigure | <del>: 4.</del> 2 | when 30% of the Primary Efficacy Analysis Population is enrolled a complete their final study visit | and |

# **List of Abbreviations**

| Abbreviation or<br>Specialized Term | Definition |
|---|---|
| ACS | acute coronary syndrome |
| ADA | anti-drug antibody |
| AE | adverse event |
| ALT | alanine transaminase |
| apoA1 | apolipoprotein A1 |
| ароВ | apolipoprotein B |
| AST | aspartate aminotransferase |
| AUC | area under the concentration-time curve |
| AUC <sub>0-∞</sub> | area under the concentration-time curve from 0 to infinity |
| AUC <sub>0-72h</sub> | area under the concentration-time curve from 0 to 72 hours |
| BP | blood pressure |
| CAD | coronary artery disease |
| CE | cholesteryl ester |
| CETP | cholesteryl ester transfer protein |
| CHD | coronary heart disease |
| C <sub>max</sub> | maximum plasma concentration |
| CMR | cardiovascular magnetic resonance |
| CTA | computed tomography angiography |
| CV | cardiovascular disease |
| ECG | electrocardiogram |
| eCRF | electronic case report form |
| EDC | electronic data capture |
| EF | ejection fraction |
| eGFR | estimated glomerular filtration rate |
| FAAN | Food and Allergy Anaphylaxis Network |
| FC | free cholesterol |
| HDL | high-density lipoprotein |
| HDL-C | high-density lipoprotein-cholesterol |
| HDL-CE | High-density lipoprotein-cholesterol ester |
| HF | heart failure |
| ICD | implantable cardioverter-defibrillator |
| ICF | informed consent form |
| ICH | International Council for Harmonisation |
| IDMC | Independent Data Monitoring Committee |
| IEC | Independent Ethics Committee |
| IRB | Institutional Review Board |
| IV | intravenous(ly) |
| IXRS | Interactive response system |

| Abbreviation or<br>Specialized Term | Definition |
|---|---|
| LAD | left anterior descending artery |
| LCAT | lecithin-cholesterol acyltransferase |
| LDL | low-density lipoprotein |
| LDL-C | low-density lipoprotein-cholesterol |
| LV | left ventricle |
| MACE | major adverse cardiac events |
| MedDRA | Medical Dictionary for Regulatory Activities |
| MI | myocardial infarction |
| MR | magnetic resonance |
| MRI | magnetic resonance imaging |
| nAb | neutralizing antibody |
| NCPV | non-calcified plaque volume |
| NO | nitric oxide |
| NOAEL | no-observed-adverse-effect-level |
| pPCI | primary percutaneous coronary intervention |
| PD | pharmacodynamics |
| PK | pharmacokinetics |
| PT | preferred term |
| RCT | reverse cholesterol transport |
| rhLCAT | recombinant human lecithin-cholesterol acyltransferase |
| SAE | serious adverse event |
| SID | subject identification |
| SOC | system organ class |
| STEMI | ST segment elevation myocardial infarction |
| sWFI | sterile water for injection |
| TEAE | treatment-emergent adverse event |
| TESAE | Treatment-emergent serious adverse event |
| TFG | TIMI flow grade |
| TIMI | Thrombolysis in Myocardial Infarction |
| ULN | upper limit of normal |
| USA | United States of America |

### 1 INTRODUCTION

This document describes the statistical analysis for protocol D5780C00007, A Randomized, Placebo controlled Phase 2b Study to Evaluate the Safety and Efficacy of MEDI6012 in Acute ST Elevation Myocardial Infarction. An overview of the study design and objectives are provided in Section 2 (pg. 6). Details for statistical methods and general conventions are provided in Section 3 (pg. 11). In addition, a set of table templates and specifications will be included in a statistical programming plan (SPP) to complement this document.

#### 2 STUDY OVERVIEW

### 2.1 Study Objectives

### 2.1.1 Primary Study Objective(s)

The primary objective and associated endpoint is presented in Table 2.1.

Table 2.1 Primary Objective and Associated Endpoint

| Type | Objective | Endpoint |
|---|---|---|
| Efficacy | To evaluate the effect of MEDI6012 | Infarct size as a percentage of LV mass measured on delayed-enhanced CMR imaging 10-12 weeks post-MI compared to placebo. |

CMR = cardiovascular magnetic resonance; LV = left ventricle; MI = myocardial infarction.

# 2.1.2 Secondary Study Objectives

Secondary objectives and associated endpoints are presented in Table 2.2.

Table 2.2 Secondary Objectives and Associated Endpoints

| Type | Objective | Endpoint(s) |
|---|---|---|
| Efficacy | To evaluate the effect of MEDI6012 on systolic function of the LV compared to placebo. | EF measured by cine MRI at 10-12 weeks post-MI compared to placebo. |
| Efficacy | To evaluate the effect of MEDI6012 on non-calcified coronary plaque regression/progression from baseline to 10-12 weeks compared with placebo. | Change in NCPV in the coronary arteries from index CTA to 10-12 weeks post-MI compared with placebo. |
| Efficacy | To evaluate the effect of MEDI6012 on remodeling of the left ventricle measured by myocardial mass and volumes. | Myocardial mass and LV volumes at end-systole and end-diastole. |
| Safety | To evaluate the safety and tolerability of MEDI6012. | Incidence of TEAEs and TESAEs. |

Table 2.2 Secondary Objectives and Associated Endpoints

| Type | Objective | Endpoint(s) |
|---|---|---|
| PK, and | To describe the PK and immunogenicity of | LCAT mass and presence of ADAs. |
| Immunogenicity | MEDI6012. | |

ADAs = anti-drug antibodies; CTA = computed tomography angiography; EF = ejection fraction; LCAT = lecithin-cholesterol acyltransferase; LV = left ventricular; MI = myocardial infarction; MRI = magnetic resonance imaging; NCPV = non-calcified plaque volume; PK = pharmacokinetic(s); TEAE = treatment-emergent adverse event; TESAE = treatment-emergent serious adverse event.

## 2.1.3 Exploratory Study Objectives

Exploratory objectives and associated endpoints are presented in Table 2.3.

Table 2.3 Exploratory Objectives and Associated Endpoints



CTA = computed tomography angiography; CV = cardiovascular; MI = myocardial infarction; pPCI = primary percutaneous coronary intervention; TFG= TIMI flow grade; TIMI = thrombolysis in myocardial infarction.

## 2.2 Study Design

This is a Phase 2b, randomized, placebo controlled- study to evaluate the efficacy, safety, pharmacokinetics/pharmacodynamics (PK/PD), and immunogenicity of repeat doses of MEDI6012 in adult subjects with acute ST segment elevation myocardial infarction (STEMI). The subject and MedImmune staff will be blinded; study sites will be trained to keep the investigator blinded. However, due to the acute nature of the study, members of the study team, and possibly the investigator, may be unblinded.



Due to the acute nature of this study, there will be a very short screening period. The study will enroll subjects presenting with acute STEMI within 6 hours of symptom onset who are planned for emergent primary percutaneous coronary intervention (pPCI). After obtaining verbal or written informed consent (as per local regulations), subjects will be assessed for eligibility, and if considered eligible, will be randomized in a 1:1 ratio into either Cohort A or Cohort B ( ). Within each cohort/dose regimen, subjects will be randomized in a 2:1 ratio to receive MEDI6012 or placebo prior to pPCI. In the event a dose regimen (Cohort A or Cohort B) is dropped at the interim analysis, subjects will be randomized in a 1:1 ratio to receive MEDI6012 or placebo for the remaining dose regimen.

Figure 2.1 Overall Study Schema



CMR = cardiovascular magnetic resonance (imaging); CTA = computed tomography angiography; D = study day; N = number of subjects; pPCI = primary percutaneous coronary intervention; STEMI = ST elevation myocardial infarction.

The study flow diagrams for Cohort A and Cohort B are presented in Figure 2.2 and Figure 2.3, respectively.



CCU = cardiac care unit; CMR = cardiovascular magnetic resonance (imaging); D = day; ED = emergency department; PCI = percutaneous coronary intervention; STEMI = ST elevation myocardial infarction.



CCU = cardiac care unit; CMR = cardiovascular magnetic resonance (imaging); CTA = computed tomography angiography; D = day; ED = emergency department; PCI = percutaneous coronary intervention; STEMI = ST elevation myocardial infarction.

## 2.3 Treatment Assignment and Blinding

An IXRS will be used for randomization to a treatment regimen. A subject will be considered randomized into the study when the investigator notifies the IXRS that the subject meets eligibility criteria. Randomization will be stratified by infarct location. Subjects will be randomized in a 1:1 ratio to one of 2 cohorts, Cohort A ( ) and Cohort B ( ). Within each dose regimen, subjects will be randomized in a 2:1 ratio to receive MEDI6012 or placebo, see Figure 2.1.

In the event that a dose regimen is dropped at the interim analysis, subjects will be randomized in a 1:1 ratio to receive MEDI6012 or placebo for the remaining dose regimen.

The randomization will be stratified by infarct location, ensuring a similar distribution of anterior vs non-anterior infarcts between the active and placebo groups. In addition, the distribution of subjects with anterior versus non-anterior MIs will be monitored over the course of the study. The goal is that > 50% of the final randomized population will be anterior MI. Therefore, the number with non-anterior MI will be monitored via the IXRS and capped by the study team.

This is a blinded study in which MEDI6012 and placebo are nearly identical in appearance. The subject/legal representative and the Sponsor will not be aware of the treatment received

(ICH E9). The unblinded individual preparing the first dose of investigational product for administration in the catheterization laboratory will be aware of the treatment received. The unblinded administrator will be trained to not reveal treatment assignment to the investigator or other clinical and study staff. The site will be asked to take reasonable steps to maintain the blind. Subsequent doses after Dose 1 will be prepared by an unblinded pharmacist. Sites are encouraged to take all reasonable steps to keep site staff involved in follow up assessments after Day 1 blinded to randomization group.

### 2.4 Sample Size



## 3 STATISTICAL METHODS

### 3.1 General Considerations

An initial database lock for the purpose of clinical study analysis and reporting will be performed when the last randomized subject completes the Day 70 to 84 visit or is discontinued prior to that visit; if no subjects are ongoing in the Extended Follow-up period, then this database lock will be considered the final database lock for the study.

If subjects are ongoing in the Extended Follow-up period, a second database lock will occur after all subjects who entered the Extended Follow-up period have completed their Week 25,

39, or 52 visits as needed or are discontinued prior to these visits, and this will be considered the final database lock. If the last Extended Follow-up visit occurs before the last Day 70 to 84 visit on the study, the second database lock will not be needed.

The study will be unblinded to the sponsor at the time of initial database lock. The site, subjects, and local CRO personnel will remain blinded to treatment assignment until the final database lock is declared.

Safety data will be generated for the Extended Follow-up period and summarized as an addendum to the clinical study report.

Data will be provided in listings sorted by treatment group and subject number. Tabular summaries will be presented by treatment group with placebo group combined when appropriate. Categorical data will be summarized by the number and percentage of subjects in each category. Continuous variables will be summarized by descriptive statistics. Baseline values will be defined as the last valid assessment prior to the first administration of investigational product on Day 1 unless data are missing, in which case, baseline will be defined as the last value prior to dosing. All statistical tests will be one-sided (based on protocol amendment) at an alpha = 0.05 significance level unless stated otherwise. Confidence intervals will be one-sided (based on protocol amendment) and nominal p-values will be reported when appropriate.

Data analyses will be conducted using the SAS® System Version 9.3 or higher (SAS Institute Inc., Cary, NC) unless otherwise specified.

# 3.2 Analysis Populations

The analysis populations are defined in Table 3.1.

Table 3.1 Analysis Populations

| Population | Description |
|---|---|
| ITT Population | The ITT Population consists of subjects who are randomized, and will be analyzed according to their randomized treatment group. |
| As-treated<br>Population | The As-treated Population consists of randomized subjects who receive any study investigational product. Subjects who receive only placebo doses will be analyzed with the placebo group; conversely, subjects who receive any dose of MEDI6012 will be analyzed with the MEDI6012 group. |
| Primary Efficacy<br>Analysis<br>Population | Randomized subjects who receive at least doses of investigational product with TFG 0 or 1 on initial angiography. Subjects who receive all placebo doses will be analyzed with the placebo group; conversely, subjects who receive doses of MEDI6012 will be analyzed with the MEDI6012 group. |

Table 3.1 Analysis Populations

| Population | Description |
|---|---|
| Efficacy Analysis<br>Population –TIMI<br>2-3 | Randomized subjects who receive at doses of investigational product with TFG 2 or 3 on initial angiography. Subjects who receive all placebo doses will be analyzed with the placebo group; conversely, subjects who receive of MEDI6012 will be analyzed with the MEDI6012 group. |
| Efficacy Analysis<br>Population TIMI –<br>0-3 | Randomized subjects who receive at of investigational product with TFG 0 to 3 on initial angiography. Subjects who receive all placebo doses will be analyzed with the placebo group; conversely, subjects who receive doses of MEDI6012 will be analyzed with the MEDI6012 group. |
| CTA Analysis<br>Population | Randomized subjects in the regimen who receive a full treatment course of investigation product. The subjects who receive placebo doses will be analyzed with the placebo group; conversely, subjects who receive dose of MEDI6012 will be analyzed with the MEDI6012 group. |
| Immunogenicity<br>Population | All subjects in the as-treated population who have at least one serum sample for immunogenicity testing. |
| PK Population | All subjects in the as-treated population who have at least one detectable serum concentration measurement for LCAT mass. |

CTA = computed tomography angiography; ITT = Intent-to-treat; LCAT = lecithin-cholesterol acyltransferase; PK = pharmacokinetic; TFG = TIMI flow grade; TIMI = Thrombolysis in Myocardial Infarction.

## 3.3 Study Subjects

## 3.3.1 Subject Disposition and Completion Status

A summary of subject eligibility and randomization as well as treatment group received (including summary of subjects randomized but not treated) will be provided. In addition, disposition of subjects throughout the study with respect to completion of treatment and follow-up will be provided.

#### 3.3.2 Demographics and Baseline Characteristics

Demographic information related to sex, age, race, ethnicity, weight, height, and body mass index will be presented by treatment group and for all subjects combined. A summary of baseline disease characteristics may include, but not be limited to medical history and acute cardiovascular disease history.

### 3.3.3 Study Drug Exposure

The number of subjects for the exposure to investigational product will be summarized descriptively by the total number of dose received.

The entire dose administered (ie, Yes vs No), the reason(s) why the subject was not administered entire dose and the reason(s) why the subject did not receive any investigational product (ie, adverse events [AEs] vs other) will be provided in the listing.

#### 3.3.4 Concomitant Medications

Concomitant medications will be coded using the latest available version of the World Health Organization Drug Dictionary and summarized by preferred term with frequency and percentage by treatment group. In addition, concomitant medications will be summarized by Anatomical Therapeutic Chemical Classification System.

## 3.4 Efficacy Analyses

### 3.4.1 Primary Efficacy Endpoint(s) and Analyses

### 3.4.1.1 Primary Efficacy Endpoint(s)

The primary efficacy endpoint is the infarct size, expressed as a percentage of LV mass measured on delayed-enhanced CMR imaging, in 10–12 weeks post- MI.

### 3.4.1.2 Handling of Dropouts and Missing Data

Missing data will not be imputed.

### 3.4.1.3 Primary Efficacy Analysis

The primary efficacy endpoint is the infarct size in 10-12 weeks post MI. The endpoint will be log-transformed due to its skewed distribution and be analyzed by means of 2-sample t-test. The treatment effect is estimated by the geometric mean ratio of MEDI6012 to placebo as well as its 95% CI. Infarct size records with zero value, will be imputed by half of the minimum of the non-zero records prior to the log transformation.

#### 3.4.1.4 Additional Analyses of the Primary Efficacy Endpoint(s)

The primary population is the primary efficacy analysis population (TIMI 0-1). Similar analysis will also be performed for the Efficacy Analysis Population with TIMI 0-3, the efficacy analysis population with TIMI 2-3, and the ITT Population.

Non-parametric (distribution-free) methods will be applied to primary endpoint data if applicable.

#### 3.4.1.5 Subgroup Analyses

The primary endpoint of infarct size will be analyzed for the following subgroups. The first set of subgroups are based on baseline characteristics and time of treatment administration.

• Sex: male vs female

- Diabetic vs non-diabetic
- Smoker vs non-smoker
- Infarct location: anterior vs non-anterior
- TIMI Flow Grade 0 vs 1 vs 2 vs 3 pre-pPCI
- TIMI Flow Grade 0 or 1 vs 2 or 3 pre-pPCI
- Above vs below the median door-to-device time
- Above vs below the median symptom onset-to-device time
- Above vs below the median symptom onset-to-door time

The second set of subgroups, outlined in Table 3.2, are based on post-randomization outcomes and will not be used to make comparisons between treatment and placebo.

Table 3.2 Post-randomization Analysis Subgroups

| Endpoint | Comparison Groups |
|---|---|
| Infarct size by culprit vessel location determined by baseline invasive coronary angiography | LAD vs Non-LAD LAD vs Left Circumflex Artery vs Right Coronary Artery |
| Infarct size by timing of drug administration | Investigational product administration before vs after pPCI Above vs below the median time between Dose 1 and pPCI |
| Infarct size by post-pPCI TIMI Flow Grade | TIMI Flow Grade 0 vs 1 vs 2 vs 3 post-pPCI TIMI Flow Grade 0 or 1 vs 2 or 3 post-pPCI |

| Infarct size by lipid and apolipoprotein | Above vs. below the median HDL at |
|---|---|
| levels | baseline |
| | Above vs. below the median HDL change from baseline |
| | Above vs. below the median apoA1 at baseline |
| | Above vs. below the median apoA1 change from baseline |
| Infarct size by cardiovascular event status | Any CV event vs no CV event |
| | HF Hospitalization vs No HF |

LAD = left anterior descending artery; pPCI = primary percutaneous coronary intervention; CV = cardiovascular; HF = heart failure

# 3.4.2 Secondary Efficacy Endpoint(s) and Analyses

### 3.4.2.1 Secondary Efficacy Endpoint(s)

Secondary efficacy endpoints include ejection fraction (EF) measured by cine MRI at 10–12 weeks post-MI, change in NCPV in the coronary arteries from index CTA to 10–12 weeks post-MI, and myocardial mass and left ventricular volumes at end-systole and end-diastole.

## 3.4.2.2 Handling of Dropouts and Missing Data

Missing data will not be imputed.

### 3.4.2.3 Secondary Efficacy Analyses

EF, myocardial mass, and left ventricular volumes will be analyzed using t-test, if appropriate, based on the Primary Efficacy Analysis Population, the Efficacy Analysis Population – TIMI 2-3; Efficacy Analysis Population – TIMI 0-3; as treated, and the ITT Population.

Change from index CTA in NCPV will be analyzed using t-test, if appropriate, based on CTA Analysis, As-treated, and ITT Populations.

Parameters will first be evaluated for normality which will be evaluated using Q-Q plots.

If the distribution appears to be normal, the endpoint will be analyzed by a 2-sample t-test. The treatment effect is estimated by difference in means of MEDI6012 to placebo as well as its 95% CI.

If the distribution appears to be log-normal, the endpoint will be log-transformed due to its skewed distribution and be analyzed by a 2-sample t-test. The treatment effect is estimated by the geometric mean ratio of MEDI6012 to placebo as well as its 95% CI.

Non-parametric (distribution-free) methods will be applied to the endpoint data if applicable.

### 3.4.2.4 Subgroup Analyses

The secondary endpoints will be analyzed for the subgroups listed below, which includes a mixture of subgroups defined before and after randomization. As for the primary efficacy endpoint, subgroups defined after randomization will not be used to make comparisons between active and placebo arms.

- Sex: male vs female
- Diabetic vs non-diabetic
- Infarct location: anterior vs non-anterior
- Infarct location: LAD vs non-LAD
- Infarct Location: LAD vs LCX vs. RCA
- TIMI Flow Grade 0 vs 1 vs 2 vs 3 pre-pPCI
- TIMI Flow Grade 0 or 1 vs 2 or 3 pre-pPCI
- TIMI Flow Grade 0 vs 1 vs 2 vs 3 post-pPCI
- TIMI Flow Grade 0 or 1 vs 2 or 3 post-pPCI
- Above vs below the median door-to-device time

- Above vs below the median symptom onset-to-device time
- Above vs below the median symptom onset-to-door time
- Drug administration before vs after pPCI
- Above vs below the median time between dose 1 and pPCI
- Above vs below the median HDL at baseline
- Above vs below the median HDL change from baseline
- Above vs below the median apoA1 at baseline
- Above vs below the median apoA1 change from baseline
- Cardiovascular Event vs No Cardiovascular Event
- HF Hospitalization vs No HF Hospitalization
- Prior statin vs statin naïve
- Baseline LDL-C  $\leq 100 \text{ vs} > 100 \text{ mg/dL}$
- Baseline LDL-C  $\leq 70 \text{ vs} > 70 \text{ mg/dL}$

### 3.4.3 Other Efficacy Analyses



#### 3.5.1.2 Analysis of Pharmacodynamic Endpoint

The PD markers measured at each time point and change from baseline at each post-baseline time point will be summarized using descriptive statistics by treatment group with placebo group combined when appropriate.

# 3.6 Safety Analyses

#### 3.6.1 Adverse Events and Serious Adverse Events

Safety analysis will be based on the As-treated Population. AE collection begins after randomization and lasts until the end of the study. SAE collection begins after the subject signs the informed consent document and lasts until the end of the study. Adverse events will be coded using the Medical Dictionary for Regulatory Activities (MedDRA) by system organ class (SOC) and preferred term (PT). Specific AEs will be counted once for each subject for calculating rates, but will be presented in total in subject listings. If the same AE occurs multiple times within a particular subject, the highest severity and level of causality will be reported. All treatment-emergent adverse events will be summarized overall and by

MedDRA SOC and PT, by severity and relationship to investigational product. In addition, summaries of deaths, serious adverse events, and treatment discontinuations due to AEs will be provided.

### 3.6.2 Adverse Events of Special Interest

Not applicable.

#### 3.6.3 Deaths and Treatment Discontinuations due to Adverse Events

Deaths, and AEs leading to discontinuation of investigational product will be summarized.

### 3.6.4 Clinical Laboratory Evaluation

Clinical laboratory safety tests including serum chemistry and hematology parameters will be summarized using descriptive statistics at each time point by treatment group with placebo group combined when appropriate. Change from baseline to each post-baseline time point in these data will also be summarized, where appropriate. A shift table will be provided for these clinical laboratory parameters where possible.

#### 3.6.4.1 Vital Signs

Vital sign results will be summarized using descriptive statistics at each time point by treatment group.

#### 3.6.4.2 Electrocardiogram

Not applicable.

# 3.7 Immunogenicity

Anti-drug antibody (ADA) incidence rate and titer will be tabulated for each treatment group. Samples confirmed positive for ADA will be tested and analyzed for neutralizing antibodies and summarized similarly.

#### 3.8 Pharmacokinetics

Serum MEDI6012 mass concentration time profiles will be summarized for MEDI6012-treated subjects by dose cohort by visit.

Additional PK analyses may be conducted as appropriate. Data obtained in this study may be pooled with other MEDI6012 studies to perform population PK analysis and/or PK/PD analysis.

## 3.9 COVID-19 Analyses

COVID-19 study disruptions may be summarized if applicable.

Additional analyses may be performed to explore the impact of COVID-19 and implemented contingency measures (eg, subjects discontinued from study treatment and/or study, protocol deviations related to COVID-19) on the safety and efficacy results reported for the study.

In addition, listings may be provided for

- subjects affected by the COVID-19 pandemic
- subjects with reported issues in the clinical trial management system due to COVID-19 pandemic

#### 4 INTERIM ANALYSIS

Two interim analyses are planned. The objectives of the first interim analysis will be to assess futility and potentially to drop a dose regimen. The analysis, which will be conducted after 30% of the Primary Efficacy Analysis Population (assumed 40% rate of exclusion from the primary efficacy analysis population is expected due to TFG 2 or 3 flow in the infarctrelated artery on initial angiography and other reasons for subsequent exclusion or drop-out) based on the original sample size (N = 74) is enrolled, will require that > 50% of subjects (N > 37) have acute anterior STEMI and have completed their final study visit. The first interim analysis will be conducted through the Independent Data Monitoring Committee (IDMC). The second interim analysis is planned to accelerate decision on future development options for MEDI6012 and will be performed once 60% of the Primary Efficacy Analysis Population (assumed 50% rate of exclusion from the primary efficacy analysis population is expected due to TFG 2 or 3 flow in the infarct-related artery on initial angiography and other reasons for subsequent exclusion or drop-out) based on the revised sample size (N = 162) is enrolled and will require that > 50% of subjects (N > 81) have acute anterior STEMI and have completed their final study visit. Details of the second interim analyses will be specified in the unblinding plan. The sponsor and Principal Investigator will monitor the statistical assumptions in a blinded fashion and schedule the interim analyses accordingly.

The assessment of futility will be based on predictive power, which is conditional power averaged over the distribution of the observed treatment effect at the time of interim analysis. The futility analysis will include all available data at the time of the interim data cut.

The predictive power based on the empirical trend observed at the interim analysis will be calculated by

predictive power 
$$pp= \Phi(rac{z_{ au}-z_{1-lpha/2}\sqrt{ au}}{\sqrt{1- au}})$$

 $\tau$  is the information fraction at the interim analysis,  $z_{\tau}$  is the observed value of the test statistic at the interim,  $\alpha$  is the two-sided significance level at the final analysis based on the original protocol, and  $\Phi$  is the standardized normal density function.

Each MEDI6012 dose regimen will be compared to the combined placebo group (pooled over dose regimens).

The study may be declared as "futile" if for both the 2-dose and the regimens the calculated predictive power is < 20% for

- infarct size in the Primary Efficacy Analysis Population; AND
- ejection fraction in the Primary Efficacy Analysis Population; AND
- infarct size in the Efficacy Analysis Population TIMI 0-3; AND
- ejection fraction in the Efficacy Analysis Population TIMI 0-3.

The regimen may be dropped if the calculated predictive power is < 20% for

- infarct size in Primary Efficacy Analysis Population; AND
- ejection fraction in Primary Efficacy Analysis Population; AND
- infarct size in Efficacy Analysis Population TIMI 0-3; AND
- ejection fraction in Efficacy Analysis Population TIMI 0-3.

For illustration purposes, Figure 4.1 provides the estimated predictive power when the observed infarct size reduction varies from -20 to 50% in the Primary Efficacy Analysis Population. The 20% predictive power translates into an infarct size reduction of approximately 7%. A value of 50% will result in 18% infarct size reduction, which is the minimally detectable treatment effect for this study. Figure 4.2 provides the estimated predictive power when the observed ejection fraction increase varies from a -5 to 10% in the

Primary Efficacy Analysis Population. Calculated predictive power will be based on observed data.

Figure 4.1 Predictive power against observed interim relative infarct size reduction when 30% of the Primary Efficacy Analysis Population is enrolled and complete their final study visit



Figure 4.2 Predictive power against observed interim ejection fraction increase when 30% of the Primary Efficacy Analysis Population is enrolled and complete their final study visit



Before declaring futility, the IDMC will evaluate data from CTA measurements for plaque regression as well as clinical efficacy endpoints (cardiovascular death, heart failure, myocardial infarction and stroke) and consider these findings in their recommendations regarding futility. If significant benefits for plaque regression and/or clinical outcomes are observed, the IDMC may recommend the data be reviewed by the sponsor's unblinded review committee (URC) for consideration to continue the trial even if the futility criteria for infarct size and ejection fraction are met. Clinical efficacy outcomes will be presented as best-available data [i.e., Clinical Events Committee (CEC) adjudicated + unadjudicated events] as well as CEC adjudicated-only data.

### 5 REFERENCES

<< Reference: Lan, Gordon K. K., Hu, Peter and Proschan, Michael A. A Conditional Power Approach to the Evaluation of Predictive Power: Statistics In Biopharmaceutical Research May 2009, Vol 1, No. 2.>>

#### 6 VERSION HISTORY

| Version | Date | Summary of Changes | Reason for Change |
|---|---|---|---|
| 1.0 | 04Jun2018 | Initial document | Initial document |
| 2.0 | 01Jul2018 | Revised the section 3.2 Analysis | Incorporated team comments. |
| First | | Populations. | |
| Approv | | -Primary Efficacy Analysis population: | If Patient gets of placebo and then |
| ed | | Subjects who receive "2" or more doses of | 1 dose of MEDI6012 at end, we won't put |
| Version | | MEDI6012 will be placed to MEDI6012 | in the MEDI arm when assessing efficacy. |
| in e- | | group. | We modified the language for the |
| TMF/V | | | clarification. Primary efficacy analysis |
| eeva | | Subjects who receive "6" doses of | population: Randomized subjects who |
| Vault | | | receive at least doses of |
| | | | investigational product with TFG 0 or 1 or |
| | | | initial angiography. Subjects who receive |
| | | Revised the section 3.4.1.5 Subgroup | all placebo doses will be included in the |
| | | Analyses. | placebo group; conversely, subjects who |
| | | - Above vs below the median symptom | receive doses of MEDI6012 will be |
| | | onset-to-"device" time | placed to MEDI6012 group. |
| | | Added section 3.6.4.2 Electrocardiogram | If Patient gets doses of placebo and then |
| | | - Electrocardiogram will be summarized | 1 dose of MEDI6012 at end, we won't put |
| | | using descriptive statistics at end of the | in MEDI arm when assessing CTA |
| | | study by treatment group. | analysis. We modified the language for |
| | | | the clarification. CTA Analysis |

| Add more details of interim analysis (e.g., predictive power). Add reference of formula of predictive power. Add data handling approach of zero infarct size. Align with protocol amendment with updated numbers related to sample size inflation and changes from two-sided to one-sided significance/alpha. Align with protocol amendment for potential 2 DBLs and extended follow-up period data report. Add statistical checking for the data distribution and applicable statistical testing based on distribution assumption to ensure the statistical appropriateness Add COVID-19 subsection and analysis Remove subgroup of statin therapy intensity Remove ECG language which is not applicable Align with protocol amendment with updated CV endpoints | | | Population: Randomization subjects in regimen who receive a full treatment course of investigation product. Subjects who receive all placebo doses will be included in the placebo group; conversely, subjects who receive of MEDI6012 will be placed to MEDI6012 group. Currently the eCRF database captures symptom onset time and device time. We changed balloon to device for subgroup analysis. We added section 3.6.4.2 for Electrocardiogram. |
|---|---|---|---|
| updated CV endpoints | 3.0 | 03Dec2020 | Add reference of formula of predictive power. Add data handling approach of zero infarct size. Align with protocol amendment with updated numbers related to sample size inflation and changes from two-sided to one-sided significance/alpha. Align with protocol amendment for potential 2 DBLs and extended follow-up period data report. Add statistical checking for the data distribution and applicable statistical testing based on distribution assumption to ensure the statistical appropriateness Add COVID-19 subsection and analysis Remove subgroup of statin therapy intensity Remove ECG language which is not applicable Align with protocol amendment with |



#### **Certificate Of Completion**

Envelope Id: 6479FDB22D46424AA9DD72933481FD02

Status: Completed

Subject: Please DocuSign: D5780C00007 Statistical Analysis Plan V3.0.docx, D5780C00007 Statistical Analy...

Source Envelope:

Document Pages: 27 Signatures: 4 Certificate Pages: 3 Initials: 0

AutoNav: Enabled

Envelopeld Stamping: Disabled

Time Zone: (UTC+01:00) Brussels, Copenhagen, Madrid, Paris

Envelope Originator:

Puerta de Hierro

Guadalajara, Jalisco 45116

IP Address: 5

#### **Record Tracking**

Status: Original

04-Dec-20 | 14:15

Holder:

Location: DocuSign

Sent: 04-Dec-20 | 14:27 Viewed: 04-Dec-20 | 14:52

Signed: 04-Dec-20 | 14:52

#### Signer Events

#### Signature

#### **Timestamp**

AstraZeneca

Security Level: Email, Account Authentication

(None)

Signature Adoption: Pre-selected Style

Using IP Address:

### **Electronic Record and Signature Disclosure:**

Accepted: 07-Feb-20 | 21:00

ID: ce7ecddc-69d8-439f-af15-78b7ffd4c7a3

Sent: 04-Dec-20 | 14:27

Viewed: 04-Dec-20 | 14:37 Signed: 04-Dec-20 | 14:37

Dr

AstraZeneca

Security Level: Email, Account Authentication

(None)

Signature Adoption: Pre-selected Style

Using IP Address:

#### **Electronic Record and Signature Disclosure:**

Accepted: 21-Feb-20 | 06:22

ID: 60f39848-df04-4f4f-b38a-07cce0c831a2

Sent: 04-Dec-20 | 14:27 Resent: 08-Dec-20 | 01:22

Viewed: 08-Dec-20 | 05:43 Signed: 08-Dec-20 | 05:44

Security Level: Email, Account Authentication

(None)

Signature Adoption: Pre-selected Style

Using IP Address:

#### **Electronic Record and Signature Disclosure:**

Accepted: 08-Dec-20 | 05:43

ID: 91f643b6-1542-4b52-958b-71097b9e9e04

AstraZeneca

(None)

Signature Adoption: Pre-selected Style

Using IP Address:

SENIOR PRINCIPAL STATISTICIAN

Security Level: Email, Account Authentication

**Electronic Record and Signature Disclosure:** 

Accepted: 31-Jan-20 | 12:53

ID: 0b9fb494-e2c5-414f-b036-da2b72e071e7

Sent: 04-Dec-20 | 14:27 Viewed: 04-Dec-20 | 14:27 Signed: 04-Dec-20 | 14:27

| In Person Signer Events | Signature | Timestamp |
|---|---|---|
| Editor Delivery Events | Status | Timestamp |
| Agent Delivery Events | Status | Timestamp |
| Intermediary Delivery Events | Status | Timestamp |
| Certified Delivery Events | Status | Timestamp |
| Carbon Copy Events | Status | Timestamp |
| Witness Events | Signature | Timestamp |
| Notary Events | Signature | Timestamp |
| Envelope Summary Events | Status | Timestamps |
| Envelope Sent Certified Delivered Signing Complete Completed | Hashed/Encrypted Security Checked Security Checked Security Checked | 04-Dec-20 14:27<br>04-Dec-20 14:27<br>04-Dec-20 14:27<br>08-Dec-20 05:44 |
| Payment Events | Ctatura | Timestamps |
| · • | Status | Timestamps |

Electronic Record and Signature Disclosure created on: 31-Jan-20 | 05:51 Parties agreed to:

I hereby consent to that AstraZeneca Worldwide https://www.astrazeneca.com may disclose personal information such as; full name, email address, and any other information you may supply on the electronic form to AstraZeneca affiliates and third party service providers throughout the world in relation to the handling and administration of the Electronic Signature Service solution. This consent relates to any electronic records or signatures associated with the electronic contract.

AstraZeneca and the third party administering this service store and process personal information that AstraZeneca collects from you for the purposes of operating the Electronic Signature Service solution.

This also applies after termination of the Agreement. Processing of your personal information will be done in accordance with applicable law.

You may request access to your personal data and withdraw agreement to this processing at any time by contacting us in writing at docusign-support@astrazeneca.com.

Personal details and electronic signatures of signatories contained in contracts cannot be removed once the contract has been executed and will remain part of such contracts until these are destroyed in accordance with applicable law and AstraZeneca internal data retention policies.